CLINICAL TRIAL: NCT00332917
Title: An Open Label SLV308 Safety Extension to Study S308.3.001 in Early PD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Erik van Leeuwen, Solvay Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S308.3.006; 2006-000858-45
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Early Stage Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — pardoprunox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pardoprunox

INTERVENTIONS:
Drug: Pardoprunox — 12-42 mg

SUMMARY:
This is a multicenter, 6 months open label safety extension study for all patients who are willing and eligible to continue from the pivotal, double-blind S308.3.001 trial

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed S308.3.001 trial

Exclusion Criteria:

* Patients with medically relevant abnormal findings (ECG, physical examination, AEs) at end of the maintenance phase (visit M6, week 24) of study S308.3.001

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety: laboratory data, adverse events, vital signs, ECG | 24 weeks

SECONDARY OUTCOMES:
UPDRS parts 1, 2 and 3, CGI-severity, CGI-improvement, PDQ-39 total score: all change from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (130):
- United States (25):
  - Site 284, Huntsville, Alabama
  - Site 274, Little Rock, Arkansas
  - Site 283, Fountain Valley, California
  - Site 277, La Jolla, California
  - Site 271, San Francisco, California
  - Site 279, Fort Lauderdale, Florida
  - Site 293, Gainsville, Florida
  - Site 282, Port Charlotte, Florida
  - Site 285, Sunrise, Florida
  - Site 273, Tampa, Florida
  - Site 290, Chicago, Illinois
  - Site 280, Kansas City, Kansas
  - Site 292, Bingham Farms, Michigan
  - Site 275, Traverse City, Michigan
  - Site 276, St Louis, Missouri
  - Site 287, St Louis, Missouri
  - Site 278, Las Vegas, Nevada
  - Site 286, Rochester, New York
  - Site 288, Ashville, North Carolina
  - Site 289, Charlotte, North Carolina
  - Site 294, Toledo, Ohio
  - Site 281, Pittsburgh, Pennsylvania
  - Site 291, Warwick, Rhode Island
  - Site 272, Houston, Texas
  - Site 270, Bennington, Vermont
- Argentina (9):
  - Site 200, Buenos Aires
  - Site 201, Buenos Aires
  - Site 202, Buenos Aires
  - Site 203, Buenos Aires
  - Site 204, Buenos Aires
  - Site 206, Buenos Aires
  - Site 208, Capital Federal, CBA
  - Site 207, Ciudad de Buenos Aires
  - Site 205, Córdoba
- Belgium (3):
  - Site 100, Brussels
  - Site 101, Genk
  - Site 102, Wilrijk
- Bulgaria (5):
  - Site 107, Plovdiv
  - Site 103, Sofia
  - Site 104, Sofia
  - Site 105, Sofia
  - Site 106, Sofia
- Canada (10):
  - Site 268, Barrie
  - Site 260, Calgary
  - Site 264, Greenfield Park
  - Site 263, Markham
  - Site 261, Ottawa
  - Site 266, Ottawa
  - Site 262, Québec
  - Site 265, Québec
  - Site 269, Saskatoon
  - Site 267, Toronto
- Chile (4):
  - Site 213, Providencia
  - Site 211, San Miguel
  - Site 210, Santiago
  - Site 212, Valdivia
- Colombia (5):
  - Site 221, Bogotá
  - Site 223, Bogotá
  - Site 224, Bogotá
  - Site 222, Cali
  - Site 220, Medellín
- Croatia (5):
  - Site 111, Rijeka
  - Site 112, Split
  - Site 110, Zagreb
  - Site 113, Zagreb
  - Site 114, Zagreb
- Finland (5):
  - Site 123, Kuopio
  - Site 122, Lappeenranta
  - Site 120, Oulun Yliopisto
  - Site 121, Tampere
  - Site 124, Turku
- India (7):
  - Site 196, Bangalore
  - Site 194, Hyderabaad
  - Site 193, Mumbai
  - Site 195, Mumbai
  - Site 199, New Delhi
  - Site 198, Thiruvananthapuram
  - Site 197, Visakhapatnam
- Israel (4):
  - Site 131, Haifa
  - Site 132, Petah Tikva
  - Site 133, Ramat Gan
  - Site 130, Tel Aviv
- Mexico (4):
  - Site 232, Aguascalientes
  - Site 230, Guadalajara - Jalisco
  - Site 231, Monterrey N.L.
  - Site 233, Tlalpan
- New Zealand (2):
  - Site 191, Christchurch
  - Site 190, Wellington South
- Peru (5):
  - Site 244, Barrios Altos-Lima
  - Site 241, La Victoria-Lima
  - Site 240, Lima
  - Site 243, San Isidro-Lima
  - Site 242, Surco-Lima
- Romania (4):
  - Site 143, Brasov
  - Site 140, Bucharest
  - Site 141, Craiova
  - Site 142, Mures
- Russia (10):
  - Site 158, Kazan'
  - Site 150, Moscow
  - Site 151, Moscow
  - Site 154, Moscow
  - Site 156, Moscow
  - Site 152, Saint Petersburg
  - Site 157, Saint Petersburg
  - Site 159, Saint Petersburg
  - Site 155, Smolensk
  - Site 153, Yaroslav
- Serbia (4):
  - Site 160, Belgrade
  - Site 161, Belgrade
  - Site 162, Belgrade
  - Site 163, Niš
- Slovakia (5):
  - Site 170, Bratislava
  - Site 171, Bratislava
  - Site 174, Levice
  - Site 173, Nitra
  - Site 172, Žilina
- South Africa (5):
  - Site 250, Cape Town
  - Site 252, Cape Town
  - Site 251, Durban
  - Site 253, Gauteng
  - Site 254, Pretoria
- Sweden (3):
  - Site 127, Gothenburg
  - Site 126, Norrköping
  - Site 125, Stockholm
- Ukraine (6):
  - Site 180, Kharkiv
  - Site 183, Kharkiv
  - Site 181, Kyiv
  - Site 182, Kyiv
  - Site 185, Lviv
  - Site 184, Vinnitsa